CLINICAL TRIAL: NCT06193018
Title: Ergonomic Effects of Using a Passive Upper Extremity Exoskeleton in Workers During Industrial Production Activities
Brief Title: Ergonomic Effects of Using a Professional Passive Exoskeleton
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: 2732
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Occupational Exposure
Keywords: Wearable devices; Electromyography; Ergonomics; Digital signal processing; Overhead work; Upper limbs supporting exoskeleton

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Work-related musculoskeletal disorders (WRMSD), multifactorial diseases that affect the working population and which can be caused and/or aggravated by work and occupational exposures, continue to Prevention interventions for these pathologies have recently made use of technological advancement, which has made external devices available for the assistance of human activities, i.e. occupational exoskeletons (EXO). Despite the suggestive potential inherent in these devices, their actual adoption in the working and industrial world is still uncertain due to the absence of evidence on their effectiveness, safety of use and appropriateness.

The use of EXO increases the user's ability to carry out manual tasks in different work contexts, lightening the perception of physical effort and promoting higher levels of safety, as well as promoting better performance. These advantages derive from the effective reduction in muscle activity that the use of EXO allows. A certain variability in the effects was referred to factors such as the type of work task, the type of exoskeleton adopted, the duration of use of the exoskeleton, as well as to individual differences and different behaviours at work.

The field studies, carried out so far in the automotive, manufacturing, logistics and agriculture sectors, are fundamental to understanding the actual effectiveness, practicality, safety and acceptance of EXO by the user.

This project contributes to the expansion of knowledge relating to the prevention of WRMSD through EXO, applying wearable sensors in a real working situation such as the textile sector, in which the female gender constitutes the majority of the workforce.

DETAILED DESCRIPTION:
The study involved the voluntary recruitment of eight workers in the sector, aged between 18 and 65, excluding those who had acute disabling pathologies or the presence of internal complications contraindicating the carrying out of activities involving the lumbar- pelvic.

Experimental part: performance of the identified work tasks (three different types, each assessed for biomechanical risk) by each worker in condition of use of EXO (EXO) and in condition of non-use (FREE). While carrying out the tasks (each with fixed frequency and duration parameters) in both conditions, workers were equipped with sensors applied on the dominant side, on the appropriate body points for the detection of electromyographic and kinematic data.

Processing of kinematic and electromyographic signals: the signals obtained from the inertial measurement unit (IMU) sensors were processed in order to quantify both the levels of muscular activity of each district analyzed and the postures adopted during the performance of the tasks.

General objective of the study was the evaluation of the effects of the use of EXO in a real working context, during repetitive activity of the upper limbs, in relation to muscular and postural commitment.

Specific objectives were:

* determine the level of muscular activity of the shoulder sectors (anterior and medial deltoid) and lumbar spine, in EXO and FREE conditions;
* determine the posture (ROM and temporal distribution of angular positions) of the sectors: shoulder, elbow, trunk in EXO and FREE conditions;
* determine the worker's perceptions regarding comfort, safety, fatigue, adaptability and usability of the device, in EXO conditions.

ELIGIBILITY:
Inclusion Criteria:

* workers of the textile sector

Exclusion Criteria:

* acute disabling pathologies or presence of internal complications contraindicating the carrying out of activities involving the lumbar- pelvic sector

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: workers at the company, on a voluntary basis
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
muscular activity of the shoulder sectors | baseline
  Electromyography root-mean-square (RMS) of the shoulder sectors (anterior and medial deltoid) and lumbar spine was determined in the EXO and in the FREE condition

CONTACTS AND LOCATIONS:
Overall Officials: Edda Capodaglio, PhD, Principal Investigator — Istituti Clinici Scientifici Maugeri SpA
Locations (4):
- Italy (4):
  - ICS Maugeri, Telese Terme, Bari
  - ICS Maugeri, Montescano, Pavia
  - ICS Maugeri, Bari
  - ICS Maugeri, Pavia